CLINICAL TRIAL: NCT01299129
Title: Functional and Morphologic Aspects of Intravitreal Triamcinolone for Uveitis-associated Cystoid Macular Edema
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marion Munk, Dr. med. univ, Medical University of Vienna
Other Study IDs: 070/2009
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Uveitis Related Cystoid Macular Edema
Keywords: Uveitis; Cystoid macular edema; microperimetry; functional visual acuity; intravitreal triamcinolone
MeSH Terms: conditions — Uveitis; Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Purpose:

To evaluate the effect of intravitreal triamcinolone acetonide (IVTA) on uveitis-associated cystoid macular edema (CME) using high resolution optical coherence tomography (SDOCT) in conjunction with thorough visual function testing.

Methods:

28 patients with uveitis-associated CME were examined before intravitreal triamcinolone injection (IVTA) (v1) and at day 1 (v2), week 1 (v3) and month 1 (v4) after injection. Retinal anatomy was evaluated using Cirrus HD-OCT (Carl Zeiss Meditec). Visual function testing consisted of assessing ETDRS distance visual acuity (VA), reading acuity and reading speed using a standardized German-language test (Radner Reading charts), contrast sensitivity using Pelli-Robson Contrast Sensitivity charts and fundus-controlled microperimetry using the MP-1 Microperimeter (Nidek). Here we utilized a cartesian grid consisting of a central locus and three concentric box-shaped stimulation areas. The changes of retinal anatomy over time were compared to the respective outcome of visual function.

ELIGIBILITY:
Inclusion Criteria:

* intraocular inflammation
* able to read
* > 18 years old

Exclusion Criteria:

* cataract
* amblyopia
* dyslexia
* already applicated intravitreal triamcinolone for current cystoid macular edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: uveitis ambulance patients of the department of ophthalmology, medical university vienna
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria